CLINICAL TRIAL: NCT05157542
Title: A Phase Ib Trial on the Safety and Feasibility of Neoadjuvant Low Dose Radiation, Chemotherapy and Durvalumab for Potentially Resectable Stage III Non-small Cell Lung Cancer (NSCLC)
Brief Title: Neoadjuvant LDRT Combined With Durvalumab in Potentially Resectable Stage III NSCLC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Juan LI, MD (Other)
Responsible Party: Sponsor-Investigator, Juan LI, MD, director of a department of medical oncology, Sichuan Cancer Hospital and Research Institute
Organization: Sichuan Cancer Hospital and Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EK2021001
Record Dates: First submitted 2021-05-24; First posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Stage III Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; Taxes; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm (Experimental): Durvalumab 1500mg, IV, Q3W, 2 cycles Albumin paclitaxel 260 mg/m2 +
  Carboplatin AUC5, IV, Q3W, 2 cycles Chemoradiotherapy(CRT):
  Cohort 1: 2 Gy in 5 Fraction
  Cohort 2: 2 Gy in 10 Fraction
  Cohort 3: 2 Gy in 15 Fraction
  Interventions: Drug: Durvalumab; Drug: nanoparticle albumin bound paclitaxel; Radiation: low dose radiation therapy

INTERVENTIONS:
Drug: Durvalumab — Day 1 and 22, 1500mg
Drug: nanoparticle albumin bound paclitaxel — Day1 and 22 nanoparticle albumin-bound paclitaxel 260 mg/m2 and carboplatin AUC 5
Radiation: low dose radiation therapy — 10 Gy in 5 fractions, 20 Gy in 10 fractions, 30 Gy in 15 fractions respectively in our three groups from Day1

SUMMARY:
Introduction: Although PACIFIC regimen definitive concurrent chemoradiotherapy (CRT) followed by Durvalumab consolidation therapy is considered the standard of care for most of stage III NSCLC patients, neoadjuvant immunotherapy combined with chemotherapy followed by surgery has shown the trend to be considered for some potentially resectable patients. The rationales for neoadjuvant treatment are tumor regression effect before surgery, early eradication of micrometastasis. Recently the investigators also find some clinical trials exploring the adding of 45 Gy in 25 fractions radiation to the combination of chemotherapy and immunotherapy neoadjuvant therapy and the investigators could see the safety is the most concern, especially the pneumonitis incidence. Low dose radiation could help control the toxicity induced by radiation and has synergic effect with immunotherapy. The aim of this phase Ib study is to assess the safety and feasibility of the combination of the concurrent low dose radiation, chemotherapy and Durvalumab neoadjuvant therapy, to explore which radiation dose is the best among our three-dose designs and evaluate if the combining neoadjuvant therapy could further improve MPR in the meantime no severe toxicities especially the grade 3-4 pneumonitis would happen.

Method: 9 eligible patients with histologically confirmed NSCLC (potentially resectable clinical stage III according to the American Joint Committee on Cancer 8th staging system) are enrolled. Patients receive Chemo (Day1 and 22 nanoparticle albumin-bound paclitaxel 260 mg/m2 and carboplatin AUC 5 ) and durvalumab (Day 1 and 22, 1500mg) and radiotherapy of 10 Gy in 5 fractions, 20 Gy in 10 fractions, 30 Gy in 15 fractions respectively in our three groups from Day1, followed by surgery. After surgery, patients are suggested to be treated with durvalumab for one year (every 4weeks, 1500 mg). The primary endpoints are safety and tolerability. The secondary endpoints are objective response rate (ORR), event-free survival EFS), overall survival (OS), pathologic complete response (pCR), and major pathologic response(MPR) in the primary tumor. biomarker analysis of PD-L1 using cancer tissue and LIPI, ctDNA using blood sample will be conducted pre-and post- neoadjuvant and post-surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 ≥ years.
2. Histological or cytological diagnosis of NSCLC by needle biopsy, and potentially resectable stage III confirmed by image logical examinations (CT, PET-CT or EBUS).
3. Eastern Cooperative Oncology Group (ECOG) performance-status score of 0 or 1.
4. Life expectancy is at least 12 weeks.
5. At least 1 measurable lesion according to RECIST 1.1.
6. With the feasibility or anticipated feasibility after neoadjuvant therapy to receive radical surgery;
7. Patients with good function of other main organs (liver, kidney, blood system, etc.):

1) ANC count ≥1.5×10^9/L, platelet count ≥100×10^9/L，hemoglobin ≥90 g/L; 2) the international standard ratio of prothrombin time (INR) and prothrombin time (PT) < 1.5 times of upper limit of normal (ULN); 3) Partial thromboplastin time (APTT) ≤1.5×ULN; 4) Total bilirubin ≤1.5×ULN; 5) Alanine aminotransferase (ALT) aspartate aminotransferase (AST) ≤2.5×ULN, or ALT and AST ≤5×ULN in the patients with liver metastatic tumor.

8. Patients with normal lung function can tolerate surgery; 9. Without systematic metastasis (including M1a, M1b and M1c); 10. The patient shall sign the Informed Consent Form.

Exclusion Criteria:

1. Participants who have received any systemic anti-cancer treatment for thymic epithelial tumor, including surgical treatment, local radiotherapy, cytotoxic drug treatment, targeted drug treatment and experimental treatment;
2. Administration of any Chinese medicine against cancer before administration of the drug;
3. Participants with other cancer within five years before the start of this study;
4. Participants with any unstable systemic disease (including active infection, uncontrolled hypertension), unstable angina pectoris, angina pectoris starting in the last three months, congestive heart failure (>= NYHA) Grade II), myocardial infarction (6 months before admission), severe arrhythmia requiring drug treatment, liver, kidney or metabolic diseases;
5. With activate or suspectable autoimmune disease, or autoimmune para cancer syndrome requiring systemic treatment;
6. Antibiotics were used to treat the infection for 4 weeks prior to the start of the trial;
7. Participants who were systemically treated with corticosteroids (prednisone or other corticosteroids >10 mg/ day) or other immunosuppressive agents within 2 weeks prior to first administration. In the absence of active autoimmune disease, inhaled or topical corticosteroids and adrenal hormone replacement therapy with a dose of less than 10 mg/ day of prednisone are permitted;
8. Participants who are allergic to the test drug or any auxiliary materials;
9. Participants with active hepatitis B, hepatitis C or HIV;
10. The vaccine was administered within 4 weeks of the start of the trial;
11. Participants who have undergone major surgery or severe trauma in other systems within 2 months before the start of this trial;
12. Pleural effusion, pericardial effusion or ascites that are not clinically controlled and require pleural puncture or abdominal puncture drainage within 2 weeks before inclusion;
13. The patients have active pia meningioma, uncontrolled or untreated brain metastases;
14. Pregnant or lactating women;
15. Participants suffering from nervous system diseases or mental diseases that cannot cooperate;
16. Participated in another therapeutic clinical study;
17. Other factors that researchers think it is not suitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2023-06-10 (Estimated); Study Completion 2023-06-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | 30 days after last dose up to 36 months
  Safety is based on evaluation of adverse events (AEs) and serious adverse events (SAEs) from the time of study drug administration through the End of Study visit. AEs and SAEs will be examined with National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v 4.03.

SECONDARY OUTCOMES:
ORR | 36 months
  Objective Response Rate determined by Response Evaluation Criteria in Solid Tumors
EFS | 36 months
  Event-free survival
MPR | 36 months
  Major pathological response rate
pCR | 36 months
  Pathological complete response rate

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Cancer Hospital, Chengdu, Sichuan, China